CLINICAL TRIAL: NCT03024476
Title: Optimization of Blood Pressure Management After Acute Ischemic Stroke and Its Prognostic Significance: Prospective, Randomized, Open, Blinded Outcome Evaluation, and Feasibility Trial
Brief Title: Optimization of Blood Pressure Management After Acute Ischemic Stroke and Its Prognostic Significance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Daiichi Sankyo Korea Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hee-Joon Bae, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1604/343
Record Dates: First submitted 2017-01-03; First posted 2017-01-18 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Ischemic Stroke; Hypertension
Keywords: behavioral intervention; prespecified medication algorithm; bluetooth-equipped sphygmomanometer
MeSH Terms: conditions — Ischemic Stroke; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive management arm (Experimental): Description:
  * Interventions in the intensive management arm consist of 1) behavioral intensification and 2) pharmacological intensification based on olmesartan
  * Participants will be given a wireless Bluetooth-equipped sphygmomanometer system, which is connected to the main server through the participants' own smartphone. Every blood pressure and heart rate measured will be encrypted and stored in the main server (Identical for both intervention and control groups).
  * Regarding behavioral intensification, an automated texting and call for breakthrough visit will be sent from the main server to encourage regular measurements of BP and maintain a desirable goad of BP.
  * Regarding pharmacological intensification, a specific algorithm for BP-lowering medication prescription will be provided to the responsible physicians by the steering committee.
  Interventions: Behavioral: Behavioral intensification; Drug: Pharmacological intensification based on olmesartan; Device: Bluetooth-equipped sphygmomanometer
- Control arm (Active Comparator): Description:
  * Other than a bluetooth-equipped sphygmomanometer, standard managements abiding by the most current guideline will be provided from the responsible physicians.
  * Participants will be given a Bluetooth-equipped sphygmomanometer, which is connected to the main server through the participants' own smartphone. Every blood pressure and heart rate measured will be encrypted and stored in the main server (Identical for both intervention and control groups).
  Interventions: Device: Bluetooth-equipped sphygmomanometer

INTERVENTIONS:
Behavioral: Behavioral intensification — Suggested algorithm for behavioral intensification:
  * If frequency of BP measurement ≤5 in a week, send a texting message
  * If frequency of BP measurement ≤3 in a week, make a telephone contact by research nurse
  * Target range of home-systolic blood pressure: 110 - 135
  * If rate of outlier exceeds 50% in a week (based on ≥5 measurements in a week), make a telephone contact by research nurse (applied at least 2 weeks after randomization). A call for breakthrough visit may be issued when clinically required (decided by the institutional investigator)
  * If frequency of BP measurement ≥ 10 in a week and frequency of outlier = 0 in a week, send a texting message to encourage and compliment on excellent BP management
  Arms: Intensive management arm
Drug: Pharmacological intensification based on olmesartan — * Study drug will be provided from the roll-in period.
  * Step I:
    * Use olmesartan 20 mg only if mean systolic blood pressure ≤150 mm Hg during the immediate past 2 days
    * Use olmesartan 40 mg if mean systolic blood pressure >150 during the immediate past 2 days
  * Step II: olmesartan 20 mg or 40 mg + amlodipine 5 mg
  * Step III: olmesartan 20 mg or 40 mg + amlodipine 10 mg
  * Step IV: olmesartan 20 mg or 40 mg + amlodipine 10 mg + hydrochlorothiazide 12.5 mg
  * If blood pressure profile showed high degree variability to evoke clinical concern, consider discontinuation of hydrochlorothiazide or reduction of olmesartan dose.
  * Use of beta-blockers is permitted if clinically indicated.
  * At each clinic visit regardless of regular or breakthrough visit, follow the pharmacological intensification rule.
  Arms: Intensive management arm
Device: Bluetooth-equipped sphygmomanometer — * Participants will be given a wireless Bluetooth-equipped sphygmomanometer system, which is connected to the main server through the participants' own smartphone. (Identical for both intervention and control groups)
  * Every blood pressure and heart rate measured will be encrypted and stored in the main server. (Identical for both intervention and control groups)

SUMMARY:
BOSS-Trial I is a phase 2 clinical trial with the following objectives;

1. to prove the feasibility of a Bluetooth-equipped sphygmomanometer system in real-world clinical practice and wireless connection to the main server;
2. to prove the feasibility of the BP management strategy, including the pre-specified BP range, BP management algorithm, and behavioral; and
3. to gather information for the phase 3 trial including BP variability indices and their potentials as a treatment guidance.

DETAILED DESCRIPTION:
* Elevated blood pressure is an established risk factor for recurrent stroke and vascular events in ischemic stroke survivors, but
* Current guideline (JNC VIII) has omitted or only partially covered a number of practical and important issues as follow;

  * When and how we measure blood pressure?
  * Is it justifiable to apply the same blood pressure threshold for office BP and home BP?
  * Should stroke survivors be treated by the same BP goal for non-stroke subjects?
  * Is it justifiable to apply the universal BP threshold for different mechanisms of ischemic stroke?
  * Is it really about only blood pressure or might it really be "beyond blood pressure?"
* Lifestyle modification should accompany all the pharmacological intervention but is usually in adequate to initiate behavioral changes.
* Frequent BP measurement at home will provide more detailed and reliable information than occasional office BP's.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke survivors within 7 days after onset
* ≥19 year-old male or female
* Medically and neurologically stabilized enough to take BP-lowering medication
* Mean systolic blood pressure ≥135 mm Hg during two days between at least 24 hours after onset and randomization (whether BP-lowering medication was prescribed or not)
* Capable of taking oral medication
* Capable of operating a wireless Bluetooth-equipped sphygmomanometer system and being expected to follow required procedures of the clinical trial
* Patients who provided written informed consent

Exclusion Criteria:

* Pregnant, puerperium ≤30 days or on breastfeeding
* enrolled in other interventional clinical trial
* Being transferred to rehabilitation center or institutionalized
* Being expected to have cerebral artery interventions within 3 months after randomization
* Known allergic reactions to olmesartan, amlodipine or hydrochlorothiazide
* Known severe hepatic disease
* Advanced kidney dysfunction requiring dialysis
* Being unlikely, in the opinion of the investigator, to comply with the clinical trial protocol or being unsuitable for any other reason.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Recruitment time to prespecified number of subjects | At 3 months after randomization
  Difference in days between recruitment of the first subject and last subject
Retention of included participants | At 3 months after randomization
  Ratio of completed subject over randomized subjects in each group
Frequencies of calls for breakthrough visit | At 3 months after randomization
  Mean and standard deviation of breakthrough visits per each patient in the intensive management group
Rate of patients who responded to the calls for breakthrough visit | At 3 months after randomization
  ratio of subjects response over the breakthrough visit calls
Control of blood pressure | At 3 months after randomization
  ratio of subjects with well-controlled BP in each group

SECONDARY OUTCOMES:
Frequency of out-of-range measurement | At 3 months after randomization
  Frequency of BP measurements out of the desirable BP range in a week
Weighted hit score of BP | At 3 months after randomization
  When two consecutive hits crossed over or below the margin of desirable BP, give 2x weight. Final score will be generated by dividing by total number of measurements
Vascular events | At 3 months after randomization
  Recurrent vascular events including recurrent stroke, myocardial infarction or vascular death
Hypotensive events | Until 3 months after randomization
  Complaint of dizzy spells, falls or low-BP related events by patients

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Joon Bae, MD.PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Seoul Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided